CLINICAL TRIAL: NCT03434522
Title: vBloc Now - A Prospective Observational Registry on the Maestro Rechargeable System (vBloc Therapy)
Brief Title: vBloc Now - Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: D01702-000
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-02

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: vBloc Maestro Rechargeable System — vBloc therapy consists of a neuromodulation device that delivers intermittent, controllable electrical blocking algorithms, to the intra-abdominal vagus nerve for the treatment of obesity.

SUMMARY:
This is a prospective, observational, case series registry which will collect information pertaining to experiences and health economics in individuals implanted with vBloc Therapy who are conjunctively using a weight management program. Subjects will be followed for 12 months after implant.

DETAILED DESCRIPTION:
The vBloc is a neuromodulation system that consists of the following implantable and external components:

* Implantable components: Two leads (including one electrode each for the anterior and posterior intra-abdominal vagal nerve trunks) are implanted laparoscopically on the intra-abdominal trunks of the vagus nerve and connected to a neuroregulator, which is implanted subcutaneously on the thoracic sidewall.
* External components: A mobile charger (MC) is connected to a non-invasive transmit coil, positioned over the implanted neuroregulator and secured in place using a transmit coil belt to charge and perform status checks on the neuroregulator. The MC is charged using an AC recharger. A laptop computer (CP) with proprietary software is used to control and upload data from the neuroregulator through the MC via the programmer cable. The CP is used by the clinician to change treatment parameters and assess battery recharging compliance. A torque wrench is used during the implant procedure to secure the leads into the neuroregulator.

Schedule of events following the baseline study visit include: implant, 2 week follow up, and 1, 3, 6, 9, and 12 month follow up visits. Enrolled subjects will also use the vBloc Achieve weight management program, which is a remote weight management counseling sessions with a registered dietitian to discuss healthy diet and exercise habits and weight loss goals.

The vBloc Now registry, together with vBloc Therapy and the vBloc Achieve weight management program, incorporates specific diets after the implant, routine remote counseling by an experienced registered dietitian, recommendations for physical activity, and tracking of weight, food intake, and fitness. The expectation is that patients participating in the vBloc Now registry, who comply with the diet and behavioral recommendations in combination with use of the Maestro device, will see an improvement in their overall health, whether it's related to weight loss, improvements in co-morbidities, or a better quality of life.

ELIGIBILITY:
Inclusion criteria

1. Signed informed consent
2. Body mass index (BMI) ≥ 40 kg/m2 to 45 kg/m2 or BMI ≥ 35 kg/m2 to 39.9 kg/m2 with one or more obesity related co-morbid conditions
3. Females or males. Note: females of child-bearing potential must have a negative urine pregnancy test at Screen and also within 14 days of implant procedure followed by physician-approved contraceptive regimen for the duration of the study period.
4. At least 18 years of age
5. Failure to respond to supervised diet/exercise program(s) in which the subject was engaged within the last five years
6. Ability to complete all study visits and procedures

Exclusion criteria

1. Patients with cirrhosis of the liver, portal hypertension, or esophageal varices.
2. Patients with a large (>5cm) symptomatic hiatal hernia
3. Patients for whom magnetic resonance imaging (MRI) is planned
4. Patients at high risk for surgical complications
5. Patients who have a permanently implanted, electrical-powered medical device or gastrointestinal device or prosthesis (e.g. pacemakers, implanted defibrillators, neurostimulators)
6. Patients for whom shortwave, microwave, or therapeutic ultrasound diathermy is planned Note: Diathermy is any treatment that uses high-frequency electromagnetic radiation, electric currents, or ultrasonic waves to produce heat in body tissues. Patients absolutely CANNOT be treated with any type of shortwave, microwave, or therapeutic ultrasound diathermy device whether or not it is used to produce heat. These treatments should not be applied anywhere on the body.
7. Current medical condition that, in the opinion of the investigator, would make the subject unfit for surgery or that would be exacerbated by intentional weight loss. Some examples include diagnosis of cancer, recent heart attack, recent stroke or serious trauma.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anyone 18 years of age and older with a BMI ≥ 40 kg/m2 to 45 kg/m2 or BMI ≥ 35 kg/m2 to 39.9 kg/m2 with one or more obesity related co-morbid conditions.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Real world experiences | 12 months following implant
  health data pertaining to weight and obesity comorbidities
Health economics | 12 months following implant
  Collecting data to examine quality of life and work productivity after implant

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sky Ridge, Lone Tree, Colorado
  - Christiana Institute of Advanced Surgery, Newark, Delaware